CLINICAL TRIAL: NCT03023215
Title: Brief Guided Relaxation for Women Undergoing Stereotactic Breast Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-1094; NCI-2017-00506 (Other: NCI CTRP)
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Meditation for Breast Biopsy
Keywords: Meditation; Breast Biopsy; Stereotactic Breast Biopsy; SBB; Guided meditation; Focused breathing; Electroencephalogram; EEG; Heart rate; HR; Questionnaires; Surveys
MeSH Terms: interventions — Meditation; Surveys and Questionnaires; Heart Rate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Guided Meditation Group (GM) (Experimental): Participants guided through 10 minutes of intervention by a mind-body specialist who will follow a standardized script prior to stereotactic breast biopsy (SBB). Mind-body specialist will also accompany participant during SBB to continue intervention.
  Electroencephalogram (EEG) activity and heart rate (HR) recorded at baseline, for 10 minutes prior to the SBB, throughout the SBB, and immediately following SBB.
  Self-report measures (anxiety and pain) assessed at baseline, immediately before, during, and after the SBB.
  Interventions: Procedure: Meditation; Procedure: Electroencephalogram; Behavioral: Questionnaires; Procedure: Heart Rate
- Focused Breathing Group (FB) (Active Comparator): Participants guided through 10 minutes of intervention by a mind-body specialist who will follow a standardized script prior to stereotactic breast biopsy (SBB). Mind-body specialist will also accompany participant during SBB to continue intervention.
  Electroencephalogram (EEG) activity and heart rate (HR) recorded at baseline, for 10 minutes prior to the SBB, throughout the SBB, and immediately following SBB.
  Self-report measures (anxiety and pain) assessed at baseline, immediately before, during, and after the SBB..
  Interventions: Procedure: Meditation; Procedure: Electroencephalogram; Behavioral: Questionnaires; Procedure: Heart Rate
- Standard of Care Group (SC) (Active Comparator): Participants listen to a 10 minute neutral-content audio clip from National Public Radio prior to stereotactic breast biopsy (SBB).
  Electroencephalogram (EEG) activity and heart rate (HR) recorded at baseline, for 10 minutes prior to the SBB, throughout the SBB, and immediately following SBB.
  Self-report measures (anxiety and pain) assessed at baseline, immediately before, during, and after the SBB.
  Interventions: Procedure: Electroencephalogram; Behavioral: Questionnaires; Procedure: Heart Rate

INTERVENTIONS:
Procedure: Meditation — Participants guided through 10 minutes of intervention by a mind-body specialist who will follow a standardized script prior to stereotactic breast biopsy (SBB). Mind-body specialist will also accompany participant during SBB to continue intervention.
  Arms: Focused Breathing Group (FB); Guided Meditation Group (GM)
Procedure: Electroencephalogram — Electroencephalogram (EEG) activity recorded at baseline, for 10 minutes prior to the SBB, throughout the SBB, and immediately following SBB.
  Other Names: EEG
Behavioral: Questionnaires — Self-report measures (anxiety and pain) assessed at baseline, immediately before, during, and after the SBB.
  Other Names: Surveys
Procedure: Heart Rate — Heart rate (HR) recorded at baseline, for 10 minutes prior to the SBB, throughout the SBB, and immediately following SBB.
  Other Names: HR

SUMMARY:
The goal of this behavioral research study is to learn if taking part in guided relaxation programs helps to reduce anxiety and pain during stereotactic breast biopsy. The study will also examine whether the guided relaxation programs change brain activity, heart rate, and blood pressure.

DETAILED DESCRIPTION:
Baseline Data Collection:

If participant chooses to take part in this study, they will be asked to fill out several questionnaires on an MD Anderson computer. Participant will be asked questions about anxiety, pain, and spirituality. The questionnaires will take about 20 minutes to complete.

Participant will have their heart rate and blood pressure taken, which will take about 3 minutes to complete. Participant will then have an electroencephalogram (EEG) done. An EEG is used to view a person's brain waves. The EEG should take about 5 minutes to complete. During the EEG, a snug cap which contains small electrodes will be placed on the head to measure the electrical patterns coming from the brain--much like the way a doctor listens to participant's heart from the surface of their skin. The EEG cap will stay on participant's head until the end of the study.

Study Groups:

After the baseline information is collected, participant will be randomly assigned (as in the role of a die) to 1 of 3 study groups: 2 relaxation training groups or a standard care group. Based on the way the study is designed, there is a 1 in 5 (or 20%) chance that participant will be assigned to the standard care group, and a 4 in 5 (or 80%) chance that participant will be assigned to one of the relaxation groups. Both relaxation groups will focus on helping participant to relax by focusing on their breath. At the end of participation, all groups will be given a 25 minute relaxation audio CD created by the MD Anderson Integrative Medicine Program.

Pre-Breast Biopsy Procedures:

Participants assigned to the relaxation groups will be guided through relaxation techniques for 10 minutes before the biopsy. Participants assigned to the third group will listen to 10 minutes of National Public Radio.

Participant's heart rate and EEG activity will be recorded during this 10-minute period of time. At the end of the 10-minute period before the breast biopsy, participant's blood pressure will be taken again and they will complete a 5 minute questionnaire about anxiety.

Breast Biopsy Procedures:

When it is time for the biopsy procedure, the research assistant will go with participant to their procedure room. In the procedure room, the research assistant will continue to monitor participant's heart rate and EEG activity throughout the biopsy time. If participant is in one of the relaxation groups, the relaxation guide will also accompany participant to the procedure room and will continue to be guided through relaxation during the biopsy procedure. If participant is in the standard care group, they will be provided with the usual breast biopsy care. Participant will be asked to talk about any anxiety and pain at several times during the procedure. Participant will also be asked to rest with their eyes closed during the biopsy procedure.

After the biopsy is finished, the research assistant will go with participant to a separate room, and they will have 5 minutes of EEG activity recorded, and their blood pressure will be taken. The EEG cap will then be removed, and participant will be asked to complete a questionnaire about their experience that will take less than 10 minutes to complete.

This is an investigational study.

Up to 85 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Women must have the ability to understand and read English, sign a written informed consent, and be willing to follow protocol requirements.
2. Women must be right hand dominant.
3. Women must be 18 years or older.

Exclusion Criteria:

1. Women who have a documented diagnosis of a formal thought disorder (e.g., schizophrenia) will be excluded from the study.
2. Women with a score of 3 or below on the Six-Item Cognitive Screener.
3. Women who plan to take benzodiazepine (e.g, alprazolam, diazepam, clonazepam, lorazepam) or beta-blocker (e.g., propranolol, atenolol) on the day of their SBB.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-10-26 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Participation and Completion Rate of Incorporating a Guided Meditation Program in Participants Undergoing Stereotactic Breast Biopsy (SBB) | 1 day
  Trial considered successful if over 50% of eligible patients participate and at least 80% of the consented patients complete the sessions and all the measures for the study.

SECONDARY OUTCOMES:
Effect of GM Compared to Focused Breathing (FB) and Standard Care (SC) Control Groups on Self-Reported Anxiety in Participants Undergoing SBB | 3-5 minute intervals throughout the SBB procedure
  Participants provide a rating from 0-10, with a rating of 0 indicating ''no anxiety'' and 10 indicating ''worst possible anxiety'' at 3-5 minute intervals throughout the SBB procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org